CLINICAL TRIAL: NCT01650844
Title: School-Based Telemedicine Enhanced Asthma Management: A Randomized Control Trial Using Novel Technology to Improve Preventive Asthma Care
Brief Title: School-Based Telemedicine Enhanced Asthma Management
Acronym: SB-TEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jill Halterman, Associate Professor of Pediatrics, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 42495
Record Dates: First submitted 2012-07-23; First posted 2012-07-26 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-08

CONDITIONS: Pediatric Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- School-based Telemedicine Enhanced Asthma Mangement Group (Experimental): We will use a web-based system to assess asthma severity or control and will send a symptom report to the child's primary care physician (PCP). Children randomized to the SB-TEAM group, will receive a telemedicine visit in the school health office at the start of the school year to provide an initial asthma assessment. The telemedicine provider will deliver brief asthma education and referrals to community resources, and will send a guideline-based preventive medication prescription electronically to a local pharmacy. The pharmacy will deliver the medications to home and school, and the school nurse will administer the medication as directly observed therapy throughout the school year. Follow-up telemedicine assessments will occur twice during the study period. These follow-up visits will focus on assessment of control, assessment of ongoing triggers or co-morbid conditions, and brief asthma education.
  Interventions: Other: School-Based Telemedicine Enhanced Asthma Management
- Enhanced Usual Care Group (Active Comparator): Children randomized to the enhanced usual care group will receive a symptom assessment using national care guidelines, a recommendation for appropriate preventive medications, and asthma education materials. We will use the web-based system to send a symptom report to the child's PCP with guideline-based recommendations for preventive care. We will provide systematic feedback to the family and providers at the same intervals as in the SB-TEAM group's telemedicine visits, by prompting providers to use care guidelines, and caregivers to schedule recommended follow-up visits with the PCP.
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Other: School-Based Telemedicine Enhanced Asthma Management
  Arms: School-based Telemedicine Enhanced Asthma Mangement Group
Other: Enhanced Usual Care
  Arms: Enhanced Usual Care Group

SUMMARY:
This project aims to improve guideline-based asthma care using enhanced communication and screening tools, telemedicine and directly observed therapy of preventive medications in city schools. Web-based screening will be used to identify children with persistent or poorly controlled asthma and to send reports to the child's primary care doctor. Children in the SB-TEAM group will receive a telemedicine asthma assessment in school and be prescribed a daily preventive asthma medication to be taken through school-based directly observed therapy. The overall aim of this study is to evaluate the use of the SB-TEAM intervention for improving guideline based care, enhancing adherence to effective preventive medications and at reducing morbidity among young urban children with asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Physician-diagnosed asthma (based on parent report)
2. Persistent asthma or poor asthma control (based on NHLBI guidelines). Any 1 of the following:

   * In past month, >2 days per week with asthma symptoms
   * >2 days per week with rescue medication use
   * >2 days per month with nighttime symptoms
   * >=2 asthma episodes during the past year that required systemic corticosteroids.
3. Age >=3 and =<10 years
4. Attending school in Rochester City School District preschools or elementary schools

Exclusion Criteria:

1. Inability to speak and understand English or Spanish
2. No access to a phone for follow-up surveys
3. Family planning to leave the district within fewer than 6 months.
4. The child having other significant medical conditions, including congenital heart disease, cystic fibrosis, or other chronic lung disease, that could interfere with the assessment of asthma-related measures.
5. Children in foster care or other situations in which consent cannot be obtained from a guardian.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2012-08; Primary Completion 2017-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Background] Halterman JS, Tajon R, Tremblay P, Fagnano M, Butz A, Perry TT, McConnochie KM. Development of School-Based Asthma Management Programs in Rochester, New York: Presented in Honor of Dr Robert Haggerty. Acad Pediatr. 2017 Aug;17(6):595-599. doi: 10.1016/j.acap.2017.04.008. Epub 2017 Apr 18. PMID 28434913
- [Background] Holderness H, Chin N, Ossip DJ, Fagnano M, Reznik M, Halterman JS. Physical activity, restrictions in activity, and body mass index among urban children with persistent asthma. Ann Allergy Asthma Immunol. 2017 Apr;118(4):433-438. doi: 10.1016/j.anai.2017.01.014. Epub 2017 Mar 6. PMID 28268134
- [Result] Halterman JS, Fagnano M, Tajon RS, Tremblay P, Wang H, Butz A, Perry TT, McConnochie KM. Effect of the School-Based Telemedicine Enhanced Asthma Management (SB-TEAM) Program on Asthma Morbidity: A Randomized Clinical Trial. JAMA Pediatr. 2018 Mar 5;172(3):e174938. doi: 10.1001/jamapediatrics.2017.4938. Epub 2018 Mar 5. PMID 29309483

RESULTS

PARTICIPANT FLOW:
Groups:
- School-based Telemedicine Enhanced Asthma Mangement Group: We will use a web-based system to assess asthma severity or control and will send a symptom report to the child's primary care physician (PCP). Children randomized to the SB-TEAM group, will receive a telemedicine visit in the school health office at the start of the school year to provide an initial asthma assessment. The telemedicine provider will deliver brief asthma education and referrals to community resources, and will send a guideline-based preventive medication prescription electronically to a local pharmacy. The pharmacy will deliver the medications to home and school, and the school nurse will administer the medication as directly observed therapy throughout the school year. Follow-up telemedicine assessments will occur twice during the study period. These follow-up visits will focus on assessment of control, assessment of ongoing triggers or co-morbid conditions, and brief asthma education.
  School-Based Telemedicine Enhanced Asthma Management
- Enhanced Usual Care Group: Children randomized to the enhanced usual care group will receive a symptom assessment using national care guidelines, a recommendation for appropriate preventive medications, and asthma education materials. We will use the web-based system to send a symptom report to the child's PCP with guideline-based recommendations for preventive care. We will provide systematic feedback to the family and providers at the same intervals as in the SB-TEAM group's telemedicine visits, by prompting providers to use care guidelines, and caregivers to schedule recommended follow-up visits with the PCP.
  Enhanced Usual Care
Period: Overall Study
Arm/Group | School-based Telemedicine Enhanced Asthma Mangement Group | Enhanced Usual Care Group
Started | 200 | 200
Completed ('Completed' indicates all participants who had data to include in the primary analysis.) | 199 | 196
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | School-based Telemedicine Enhanced Asthma Mangement Group | Enhanced Usual Care Group | Total
Number analyzed (Participants) | 200 | 200 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.7 (1.7) | 7.9 (1.7) | 7.8 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 76 | 153
  Male | 123 | 124 | 247
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 112 | 118 | 230
  Hispanic | 67 | 60 | 127
  Other | 21 | 22 | 43
Region of Enrollment [Number; unit: participants]
  United States | 200 | 200 | 400
Symptom-Free Days over two weeks [Mean (Standard Deviation); unit: Days] | 7.0 (5.2) | 7.4 (5.1) | 7.2 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Days Without Asthma Symptoms (Symptom Free Days)
Description: The primary outcome measure is asthma morbidity between groups. We will measure asthma morbidity by looking at the average number of days without asthma symptoms (symptom free days) over 2 weeks, during each follow-up assessment during the peak winter season (November-March). Symptom free days are defined as 24 hour periods of no asthma symptoms including, coughing, wheezing, tightness in the chest or shortness of breath. The number of symptom free days will be reported by the child's caregiver.
Time Frame: Average number of days, over 2 weeks, during peak winter season (November-March), assessed over 4 years.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | School-based Telemedicine Enhanced Asthma Mangement Group | Enhanced Usual Care Group
Number analyzed (Participants) | 199 | 196
Days | 11.6 (2.7) | 10.97 (3.2)
Statistical Analysis 1: Comparison: School-based Telemedicine Enhanced Asthma Mangement Group vs Enhanced Usual Care Group; Test type: Other — We estimated the power to detect the smallest clinically significant difference in mean SFDs post intervention between the groups, accounting for repeated measures. A sample of 400 obtains greater than 90% power to detect a difference of 0.8 SFD per 2 weeks or greater. Analyses were multivariable modified intention to treat, including all participants with post intervention data. Generalized estimating equation (GEE) models were fitted with repeated asthma outcomes; p < 0.05, Regression, Linear — Analyses were multivariable modified intention to treat, including all participants with post intervention data. Generalized estimating equation (GEE) models were fitted with repeated asthma outcomes; Mean Difference (Net) = 0.8, Standard Deviation 2.8

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | School-based Telemedicine Enhanced Asthma Mangement Group | Enhanced Usual Care Group
All-Cause Mortality (participants affected / at risk) | 0/200 | 0/200
Serious Adverse Events (participants affected / at risk) | 0/200 | 0/200
Other Adverse Events (participants affected / at risk) | 0/200 | 0/200

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT01650844/Prot_SAP_001.pdf